CLINICAL TRIAL: NCT04282564
Title: Improvement of Executive Functions With the CO-OP Method in the Adult Subject After Stroke
Acronym: FéCO-OPSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID lockdown + financial problems + no inclusion since lockdown
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0448
Record Dates: First submitted 2020-02-14; First posted 2020-02-24 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Cerebrovascular Accident
Keywords: CO-OP; executive functions; stroke; single-case experimental designs; transfer of knowledge; sens of self efficacy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CO-OP Arm (early phase A) (Experimental): Patients will be integrated during the traditional day hospitalization follow-up, at the rate of 3 sessions per week. The patient will have 2 phases : phase A: CO-OP treatment during 6 week and phase B : without specific treatment during 3 weeks.
  Interventions: Other: Co-OP treatment
- CO-OP Arm (mid phase A) (Experimental): Patients will be integrated during the traditional day hospitalization follow-up, at the rate of 3 sessions per week. The patient will have 2 phases : phase A: CO-OP treatment during 6 week and phase B : without specific treatment during 2.5 weeks.
  Interventions: Other: Co-OP treatment
- CO-OP Arm (late phase A) (Experimental): Patients will be integrated during the traditional day hospitalization follow-up, at the rate of 3 sessions per week. The patient will have 2 phases : phase A: CO-OP treatment during 6 week and phase B : without specific treatment during 2 weeks.
  Interventions: Other: Co-OP treatment

INTERVENTIONS:
Other: Co-OP treatment — The Cognitive Orientation to daily Occupational Performance (CO-OP) approach is described as "a patient-centred, performance-oriented approach to activities and problem solving that allows skills to be acquired through a process of strategy use and guided discovery". The CO-OP protocol is composed of seven key characteristics: i) the goals chosen by the patient, ii) dynamic performance analysis, iii) the use of cognitive strategies, iv) guided discovery, v) the principles of empowerment, vi) the involvement of a relative, vii) the structure of the intervention (Polatajko and Mandich, 2004/2017). CO-OP is an evidence-based approach to intervention, including evidence of its effectiveness on a physical, cognitive and emotional dimension in adults with stroke

SUMMARY:
The research focuses on top-down intervention approaches and more specifically on the Cognitive Orientation to daily Occupational Performance (CO-OP) method in the rehabilitation of executive function disorders in adult post-stroke subjects in chronic phase. The main objective of this study is therefore to improve performance in significant activities of daily living for people with chronic post-stroke dysexecutive disorders.

DETAILED DESCRIPTION:
Today, approaches to intervention with adults after stroke can be categorized into two groups: bottom-up approaches (neurodevelopmental, sensory integration, mental imagery, cognitive stimulation, perceptual-motor/kinesthetic training...) and top-down approaches (task-oriented approach, neuromotor task training, occupational performance coaching, the CO-OP approach). Although bottom-up intervention approaches have existed for several years longer than top-down approaches, in general, top-down intervention approaches have shown better results.

In the latest work with post-stroke adults with objective cognitive impairment, the data indicate the relevance of CO-OP in improving performance and satisfaction, attention, inhibition and flexibility or apathy.

This study aims to demonstrate the effectiveness of the CO-OP approach in adult post-stroke patients in chronic phase, specifically on planning function, through the Single Case Experimental Design methodology by randomized intervention (3 patients) over 6 weeks of treatment and 10 weeks of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Stroke responsible for a dysexecutive syndrome authenticated by the GREFEX battery
* Stroke more than 6 months old (chronic phase)
* Social security affiliation
* Signing of a free and informed consent following clear and detailed information.

Exclusion Criteria:

* Disorder of comprehension objectified by the - LAnguage Screening Test (LAST) (minimum score 4/8 in expression and 6/7 in comprehension)
* Significant anosognosia of dysexecutive syndrome
* Pregnant women
* Neurological condition other than stroke or psychiatric disorder
* Patient following a rehabilitation with a liberal therapist targeting executive functions during the period of participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Improved performance in significant activities of daily living | 10 weeks
  Improved performance in significant activities of daily living will be measured bi-weekly by the Canadian Occupational Performance Measurement. The score is between 1 to 10
Improved performance in significant activities of daily living | 10 weeks
  Improved performance in significant activities of daily living will be measured bi-weekly by the Performance Quality Rating Scale. The score is between 1 to 10

SECONDARY OUTCOMES:
improvement in the sense of personal effectiveness | 10 weeks
  The improvement in the sense of personal effectiveness will be measured by New General Self-Efficacy Scale (8 questions with response to 1 for strongly disagree to 5 for strongly agree)
Analytically measure of executive functions | 10 weeks
  The analytical improvement of executive functions will be measured by the Trail Making Tes
Analytically measure of executive functions | 10 weeks
  The analytical improvement of executive functions will be measured by the number span (WAIS IV)
Analytically measure of executive functions | 10 weeks
  The analytical improvement of executive functions will be measured by the Stroop test
Analytically measure of executive functions | 10 weeks
  The analytical improvement of executive functions will be measured by the test "the Tower of London"
Analytically measure of executive functions | 10 weeks
  The analytical improvement of executive functions will be measured by the Wisconsin Card Sorting test

CONTACTS AND LOCATIONS:
Overall Officials: Xavier De Boissezon, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No